CLINICAL TRIAL: NCT05159739
Title: Genetic Susceptibility to Periprosthetic Joint Infections of the Hip and Knee
Brief Title: Genetic Susceptibility to Periprosthetic Joint Infections
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Jeremy Gililland, Principle Investigator, University of Utah
Other Study IDs: 95940
Record Dates: First submitted 2021-12-02; First posted 2021-12-16 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Total Joint Arthroplasty; Periprosthetic Joint Infections
Keywords: total joint arthroplasty; periprosthetic joint infections; genetic susceptibility
MeSH Terms: conditions — Genetic Predisposition to Disease | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Draw or Saliva/Cheek Cell Sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Total Joint Arthroplasty (TJA): Recruitment of families with an increased incidence of TJI with PJI.
  Interventions: Genetic: Blood Draw or Saliva/Cheek Cell Sample:

INTERVENTIONS:
Genetic: Blood Draw or Saliva/Cheek Cell Sample: — Collected samples will immediately undergo genetic analysis to determine the presence or absence of potential candidate genes responsible for the increased incidence of PJI.
  Other Names: Genetic sample

SUMMARY:
The investigators primary objective is to identify genetic factors that may increase the risk of patients developing a periprosthetic joint infections (PJI) following total joint arthroplasty (TJA). The investigators hope that by identifying genetic predispositions we will be able to provide patient specific care pathways to prevent or minimize the risk for PJI.

DETAILED DESCRIPTION:
Surgical site infections (SSI), and more specifically periprosthetic joint infections (PJI), have plagued the orthopaedic surgeon since the introduction of total joint arthroplasty (TJA) procedures of the hip or knee in the mid twentieth century. It is estimated that the economic burden of PJI in the United States will approach 1.62 billion USD by 2020. Though methods of infection control have improved, the rate of PJI appears to have plateaued in the last several decades. Early rates of PJI in the first two decades of THA have been reported between 1 - 9%. Since the 1980's studies have reported rates between 1% - 3%. It has been suggested that as orthopaedic surgeons, doctors should not be satisfied with deep infection rates greater than 1%. Therefore, more must be done in order to prevent, or diminish the frequency, of PJI and its devastating effects on this patient population.

In hopes of allowing for early targeted prevention in potentially high-risk patients, risk calculators have been developed to identify patients at greater risk for developing infection following TJA. However, some investigators suggest that these scoring systems may not be ready for primetime use. Thus, further research is needed to improve the ability to accurately identify individuals at high risk for infection. Unfortunately, the ability to perform large scale longitudinal cohort studies needed to create and test these risk calculators isn't feasible. Thus, other methods of early identification are needed.

Genetic susceptibility testing for identifying patients at risk for disease is becoming more popular and may be a means by which patients at high-risk for PJI can be identified. A recent dermatological study on genetic risk factors for infection suggest that host attributes may play a role in the ability of the individual to be infected. When evaluating the risk of subsequent different site infection in patients with multiple TJA's, investigators suggest that some patients may be at greater risk for infection due to possible subclinical immune deficiencies. In 2013, one investigator reported familial susceptibility to surgical site infections (SSI), including but not isolated to PJI, through a large population based study. Further, a recent publication from this investigating institution demonstrated familial clustering in patients who suffered a PJI, showing an increased risk of PJI following TJA in relatives of patients who have experienced PJI. These families demonstrated infection rates of 9 - 17%. After performing a systematic review on the genetic susceptibility to PJI, the investigators concluded that though evidence exists supporting a genetic role in PJI, no definitive conclusions can be made given the relatively small amount of data available in the existing literature. The investigators further emphasize the need for prospective studies to validate previous findings and the relationship between genetic factors and PJI.

Given the evidence in the literature, the investigators hypothesize that a large familial study will provide greater evidence of a genetic susceptibility. The results of this study could validate previous research with smaller sample sizes and allow for early identification of high-risk patients via genetic susceptibility testing.

ELIGIBILITY:
Inclusion Criteria:

* Families/pedigrees which demonstrate a high-risk for PJI
* Unaffected family members, up to 3rd degree

Exclusion Criteria:

* None

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Family members (affected and unaffected) with an increased incidence of TJI with PJI.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-03-07 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Genotyping | DNA extraction and analysis will be performed immediately after collection of blood draw or saliva/cheek cell sample by a certified core lab
  Samples will undergo genetic testing to determine the presence or absence of potential candidate genes responsible for the increased incidence of PJI.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Gililland, M.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah Orthopaedic Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No